CLINICAL TRIAL: NCT02774967
Title: Comparation Between Two Surgical Techniques With Acellular Dermal Matrix in Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, professor of periodontics department, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 35907314.8.0000.5419
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Gingival Recession; Gingival Diseases; Mouth Diseases; Periodontal Atrophy; Periodontal Diseases; Stomatognathic Diseases
Keywords: root coverage; gingival recession; periodontal surgery
MeSH Terms: conditions — Gingival Recession; Gingival Diseases; Mouth Diseases; Periodontal Atrophy; Periodontal Diseases; Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- extended flap technique (Active Comparator): root coverage comparing two techniques The aim of this study was to compare and show the benefits of the extended flap technique compared to Tunnel technique both techniques using the acellular dermal matrix for root coverage.
  Other Names:
  acellular dermal matrix extended flap technique
  Interventions: Procedure: root coverage
- tunnel technique (Experimental): root coverage comparing two techniques The aim of this study was to compare and show the benefits of the extended flap technique compared to Tunnel technique both techniques using the acellular dermal matrix for root coverage.
  Other Names:
  acellular dermal matrix extended flap technique
  Interventions: Procedure: root coverage

INTERVENTIONS:
Procedure: root coverage — Root coverage with acellular dermal matrix using two techniques: advanced positional flap ou tunneling,

SUMMARY:
The gold standard for the treatment of gingival recession, is the coronal repositioning of the flap associated with the subepithelial connective tissue graft. The acellular dermal matrix (ADM) has been used as a substitute a subepithelial connective tissue graft in periodontal plastic surgery and mucogengivais, and has achieved similar results. The use of ADM has the advantage of avoiding possible pre and postoperative complications, as well as overcome the limitations presented by autograft. The different surgical techniques used for root coverage seek predictability and success. For this, besides the type of incision placements flap and graft are of utmost importance because the healing benefit and outcome.

The aim of this study is to compare two surgical techniques for root coverage and evaluate which one provides better cosmetic results and less morbidity . 20 adults , nonsmoking patients , showing multiple bilateral gingival recessions , class I or II Miller located in canine, first and second premolars are selected. Both techniques use the ADM as a graft. However , in one Quadrant partial flap will be held together with relaxing incisions through an incision intrasucular , ADM will be positioned 1 mm apical to the cementoenamel junction (CEJ) and the flap will be positioned 1 mm coronal CEJ. In the opposite quadrant a minimally invasive technique periosteal envelope above does not use relaxing incisions , preserves the buds will be held , as well as avoiding any scars, the graft will be used to ADM. The clinical parameters (probing depth, clinical attachment level, bleeding on probing index, height and width of the gingival retraction and height and thickness of keratinized gingiva) will be evaluated 2 weeks after the basic periodontal therapy and after 6 and 12 months to surgical procedures. In addition, measurements of photographic gingival recession with the aid of software will be performed.

ELIGIBILITY:
Inclusion Criteria:

ages 18 to 50 years old bilateral multiple gingival recession type Miller class I or II with at least one tooth with 3 mm in height and less than 3mm of keratinized tissue in canine and pre-molar teeth

Exclusion Criteria:

diabetics pregnant women chronic use of medication periodontitis smokings

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comparing changes for Root coverage measure (in millimeter) from baseline at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: arthur b novaes jr, PhD, Principal Investigator — FORP-USP; gabriel f bastos, MSD Student, Principal Investigator — FORP-USP
Locations (1):
- Gabriel F Bastos, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No